CLINICAL TRIAL: NCT05343338
Title: A Randomized Controlled Study of Sivelestat Sodium in Improving Pulmonary Insufficiency After Aortic Dissection Arch Surgery Under Hypothermic Circulatory Arrest
Brief Title: Improvement of Pulmonary Insufficiency After Aortic Dissection With Sivelestat Sodium
Acronym: IPIADSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2021CRF-017
Record Dates: First submitted 2022-04-10; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Aortic Dissection; Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Aortic Dissection; Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sivelestat sodium on the basis of the original treatment (Experimental): In the perioperative period, sivelestat sodium was added, and on the basis of not terminating and changing the original treatment plans.
  Interventions: Drug: Sivelestat sodium
- the original treatment (No Intervention): Only accept the original clinical diagnosis and treatment and clinical management.

INTERVENTIONS:
Drug: Sivelestat sodium — After dissolving sivelestat sodium with 0.9% sodium chloride injection, dilute the 1-day dose (4.8 mg/kg) with 50 mL of 0.9% sodium chloride injection and continue intravenously at a rate of 0.2 mg/kg/h for administration. The start time of administration was after induction of anesthesia, and at the same time, the extracorporeal circulation circuit is prefilled with 100 mg. The end time is 48 hours after admission to the ICU.
  Arms: sivelestat sodium on the basis of the original treatment

SUMMARY:
Aortic dissection (AD) is one of the most dangerous cardiovascular emergencies, with rapid onset, rapid progression, high fatality rate, and a variety of life-threatening complications. Acute lung injury (ALI) caused by AD is an important cause of many adverse outcomes. Studies have confirmed that 34.9% to 53.8% of AAD patients have ALI before surgery, and Impaired preoperative lung function may lead to worse oxygenation after AD surgery. The pathophysiological mechanism of AD-induced ALI is complex. A variety of preoperative and intraoperative risk factors can induce or aggravate ALI, such as ischemia-reperfusion injury, deep hypothermic circulatory arrest, and inflammatory reactions. At present, the clinical use of improved surgery, cardiopulmonary bypass perfusion, early anti-inflammatory treatment, and protective lung ventilation can reduce and improve perioperative ALI to a certain extent, but it is still not ideal. In recent years, inhibition of neutrophil activation and aggregation, and reduction of neutrophil elastase activity as targets for the treatment of inflammatory injury have also become an important clinical treatment measure, in order to further reduce the body's inflammatory response to improve and alleviate ALI. Sivelestat sodium, as a neutrophil elastase inhibitor, is the only approved therapeutic drug for ALI/ acute respiratory distress syndrome (ARDS) in the world. It is precisely by reducing the inflammatory infiltration of neutrophils and inhibiting neutrophil elastase activity, thereby exerting a certain protective effect on the lungs. The study takes patients with AD surgery as the research object. On the basis of not terminating and changing the original treatment plans, sivelestat sodium was added in the perioperative period to observe the incidence, and severity of ALI/ARDS in the perioperative period. It aims to explore the efficacy and safety of sivelestat sodium in the treatment of pulmonary insufficiency after AD arch surgery under hypothermic circulatory arrest.

DETAILED DESCRIPTION:
The study is a single-center, randomized, open-label, blank-controlled study, and designs to recruit AD perioperative patients admitted to the Cardiovascular Surgery Department of the First Affiliated Hospital of Xi'an Jiaotong University, between January 1, 2022 and December 31, 2022, with a total of 168 cases. After the patients who met the inclusion and exclusion criteria signed the informed consent, they were randomly assigned to the experimental group and the control group at a 1:1 ratio, with 84 cases in each group. The experimental group is additionally given sivelestat sodium in the perioperative period on the basis of the original treatment. The study was divided into two phases, the screening phase and the treatment phase. The screening period was from admission to the day of surgery to determine whether patients were suitable for the study. The treatment period is from the induction of anesthesia to the day of being transferred out from the ICU. It is necessary to complete the detailed treatment plan, and drug dosage, intraoperative and postoperative serological examinations, imaging examinations, and the patient's mechanical ventilation and oxygenation index data. Sivelestat sodium was used during and after operation in the experimental group, and the end time of administration was 96 hours after admission to the ICU. During the treatment with sivelestat sodium, the patient's original treatment plan will not be terminated or affected. The control group only received the original clinical diagnosis and treatment and clinical management. Study endpoints were defined as the day of ICU transfer, follow-up until discharge, or discontinuation/termination during the study period, or patient withdrawal from the study for any reason. During the study period, doctors will provide supportive treatment according to clinical indications, medication instructions and specifications. In the event of an adverse event, the doctor may make adjustments to the medication dose and treatment duration. The main observation indicators were the incidence of moderate to severe respiratory insufficiency (PaO2/FiO2 ≤ 200mmHg) at 24, 72, and 120 hours after surgery, on the day of transfer out of ICU, and discharge. The efficacy and safety of the drug were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 70 years old;
* Patients undergoing aortic dissection arch surgery under hypothermic circulatory arrest;
* Weight from 45 to 90kg;
* ASA cardiac function class from II to IV;
* Patients who can understand and comply with the requirements of the protocol and volunteer to participate.

Exclusion Criteria:

* Patients participating in other clinical studies;
* Patients with serious lack of medical data;
* Women who are pregnant or may become pregnant or breastfeeding;
* Patients with severe lung diseases, such as end-stage chronic obstructive pulmonary disease, chronic interstitial lung disease, etc.;
* Patients with malignant tumors;
* Preoperative oxygenation index PaO2/FiO2≤200mmHg;
* Patients with EUROScoreII mortality risk < 3%;
* Patients with APACHE II score ≥ 21;
* Patients who are judged by the researchers to be unsuitable for inclusion, such as those with mental illnesses.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2022-04-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of respiratory insufficiency | 24 hours after surgery
  Incidence of postoperative moderate to severe respiratory insufficiency (PaO2/FiO2 ≤ 200mmHg).
Incidence of respiratory insufficiency | 72 hours after surgery
  Incidence of postoperative moderate to severe respiratory insufficiency (PaO2/FiO2 ≤ 200mmHg).
Incidence of respiratory insufficiency | 120 hours after surgery
  Incidence of postoperative moderate to severe respiratory insufficiency (PaO2/FiO2 ≤ 200mmHg).

SECONDARY OUTCOMES:
Incidence of prolonged mechanical ventilation | 120 hours after surgery
  Mechanical ventilation time > 72h
Levels of neutrophil elastase activity | 24 hours after surgery
  Preoperative and postoperative blood neutrophil elastase activity levels.
Levels of neutrophil elastase activity | 72 hours after surgery
  Preoperative and postoperative blood neutrophil elastase activity levels.
Levels of neutrophil elastase activity | Date of discharge from Cardiovascular Surgery ICU for any reason, or assessed up to 4 weeks
  Preoperative and postoperative blood neutrophil elastase activity levels.
White blood cell count | 24 hours after surgery
  Blood routine examination WBC count
White blood cell count | Date of discharge from Cardiovascular Surgery ICU for any reason, or assessed up to 4 weeks
  Blood routine examination WBC count
plasma C-reactive protein | 24 hours after surgery
  serial plasma high-sensitivity CRP
plasma C-reactive protein | Date of discharge from Cardiovascular Surgery ICU for any reason, or assessed up to 4 weeks
  serial plasma high-sensitivity CRP
serum procalcitonin | 24 hours after surgery
  Serum PCT level
serum procalcitonin | Date of discharge from Cardiovascular Surgery ICU for any reason, or assessed up to 4 weeks
  Serum PCT level
serum interleukin-6 | 24 hours after surgery
  Serum IL-6 level
serum interleukin-6 | Date of discharge from Cardiovascular Surgery ICU for any reason, or assessed up to 4 weeks
  Serum IL-6 level

CONTACTS AND LOCATIONS:
Overall Officials: Tao Shi, PhD, Study Chair — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided